CLINICAL TRIAL: NCT03104621
Title: Efficacy and Tolerability of Preservative-free 0.0015% Tafluprost in Glaucoma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Gong Je Seong, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3-2013-0042
Record Dates: First submitted 2017-03-13; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Primary Open-angle Glaucoma
Keywords: preservative-free, tafluprost
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Benzalkonium Compounds; tafluprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators, patients and other study participants were blinded to treatment assignment throughout the study. Evaluator of IOP was also masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1, for the first 6 months, the subjects of group 1 used non-preservative disposable 0.0015% tafluprost product(Taflotan-S®) and then changed to 0.001% Benzalkonium chloride (BAK), 0.0015% tafluprost product (Taflotan®)for 6 months.
  Interventions: Drug: Benzalkonium chloride (BAK); Drug: 0.0015% tafluprost
- Group 2 (Experimental): Group 2, for the first 6 months, the subjects of group 2 used 0.001% Benzalkonium chloride (BAK), 0.0015% tafluprost product(Taflotan®) and then changed to non-preservative disposable 0.0015% tafluprost product(Taflotan-S®) for 6 months.
  Interventions: Drug: Benzalkonium chloride (BAK); Drug: 0.0015% tafluprost

INTERVENTIONS:
Drug: Benzalkonium chloride (BAK) — Benzalkonium chloride (BAK) is the most used preservative and is excellent for safety and stability of drug. However, it causes dry eye, corneal oedema, corneal erosion, and corneal toxicities, thus lowering the long-term tolerability for patients. A critical component when managing glaucoma patients is ensuring compliance.
Drug: 0.0015% tafluprost — Tafluprost (trade names Taflotan or Taflotan-S by Santen Pharmaceutical) is a prostaglandin analogue. It is used topically (as eye drops) to control the progression of open-angle glaucoma and in the management of ocular hypertension. In this study, tafluprost was used in all experimental group with equally concentration(0.0015%), only measured whether BAK was included or not.

SUMMARY:
The aim of this work is to evaluate efficacy and tolerability of preservative containing 0.0015% tafluprost and preservative-free 0.0015% tafluprost. Both preservative containing and preservative-free 0.0015% tafluprost will reduce intraocular pressure significantly. In addition, preservative-free 0.0015% tafluprost might improve tolerability of glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Primary open angle glaucoma and normotensive glaucoma patients who came to the outpatient clinic for regular glaucoma check-ups were enrolled.
* 2. Glaucoma was defined as the patients who had open angle confirmed by gonioscopy, optic nerve cupping (a vertical cup-disc ratio of >0.6) and or notching of the neuroretinal rim and or retinal nerve fiber defects characteristics of glaucoma, and visual field defect(i.e., a glaucoma hemi-filed test result outside normal limits, a pattern standard deviation probability of <5%, or a cluster of three or more non-edge points in location typical of glaucoma, all of which were depressed on a pattern deviation plot at a P level of <5%, and at least one of which was depressed at a P level of <1% on two consecutive visual field tests).
* 3. Normal tension glaucoma included criteria: repeated measurements of untreated IOP values of < 21mmHg. Primary open angle glaucoma included criteria: repeated measurements of untreated IOP values of ≥ 22mmHg.

Exclusion Criteria:

* 1. Phakic and pseudophakic eyes.
* 2. eyes that had been taken vitrectomy, trabeculectomy, or surgery influenced IOP

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The change of corneal erosion grade by preservative free 0.0015% tafluprost | after 1, 3, and 6 months using drug in group 1/ after 7, 9, and 12 months using drug in group 2
  Corneal erosion scales were scored according to the area of erosion. Little to no erosion was "0", erosion on 1/3 of the area of the entire cornea was "1", erosion on 2/3 of the area of the entire cornea was "2", and erosion on the entire cornea was "3"
The change of tear break up time by preservative free 0.0015% tafluprost | after 1, 3, and 6 months using drug in group 1/ after 7, 9, and 12 months using drug in group 2
  Tear breakup time was checked by slit lamp exam under corneal fluorescein dye. We asked patients not to blink, and the time was counted until tear film was torn apart (seconds)
The change of Schirmer test by preservative free 0.0015% tafluprost | after 1, 3, and 6 months using drug in group 1/ after 7, 9, and 12 months using drug in group 2
  For tear secretion, schirmer test paper was placed into the conjunctival sac at the point of 1/3 from lateral canthus under topical anaesthesia (5% Proparacaine HCl, Alcaine®, Alcon Laboratories Inc., TX, USA). After 5 minutes, we checked the wet height with tear (mm)
The change of corneal erosion grade by preservative contained 0.0015% tafluprost | after 1, 3, and 6 months using drug in group 2/ after 7, 9, and 12 months using drug in group 1
  Corneal erosion scales were scored according to the area of erosion. Little to no erosion was "0", erosion on 1/3 of the area of the entire cornea was "1", erosion on 2/3 of the area of the entire cornea was "2", and erosion on the entire cornea was "3"
The change of tear break up time by preservative contained 0.0015% tafluprost | after 1, 3, and 6 months using drug in group 2/ after 7, 9, and 12 months using drug in group 1
  Tear breakup time was checked by slit lamp exam under corneal fluorescein dye. We asked patients not to blink, and the time was counted until tear film was torn apart (seconds)
The change of Schirmer test by preservative contained 0.0015% tafluprost | after 1, 3, and 6 months using drug in group 2/ after 7, 9, and 12 months using drug in group 1
  or tear secretion, schirmer test paper was placed into the conjunctival sac at the point of 1/3 from lateral canthus under topical anaesthesia (5% Proparacaine HCl, Alcaine®, Alcon Laboratories Inc., TX, USA). After 5 minutes, we checked the wet height with tear (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Gong Je Seong, Principal Investigator — Gangnam Severance Hospital

REFERENCES:
- [Derived] Lee W, Lee S, Bae H, Kim CY, Seong GJ. Efficacy and tolerability of preservative-free 0.0015% tafluprost in glaucoma patients: a prospective crossover study. BMC Ophthalmol. 2017 Apr 28;17(1):61. doi: 10.1186/s12886-017-0453-z. PMID 28454526